Scientific title

Application of 3D magnetic resonance neurogram sequences for evaluation of Intraparotid facial nerves in patients with parotid neoplasm

## **Informed consent form in English**

Version 2

Date: 9 June 2022

NCT Number: NCT05296109



## Department of Imaging and Interventional Radiology

## The Chinese University of Hong Kong

## **Consent Form**

Title: Application of three-dimensional Resonance Neurogram Sequences for evaluation of intra-parotid facial nerves in Patients with Parotid Neoplasms

Principal Investigator: Dr. HS Leung

Co-Investigators: Dr. Jill Abrigo, Prof. Winnie CW Chu, Dr. Eric HL Lau, Dr. Ronald Lai, Dr. SM Yu, Dr. KT Wong, Prof. Ann D. King

I declare that my participation in this study is entirely voluntary:

- 1. I fully understand and voluntarily join the research study.
- 2. I have already read the information sheet of this study and fully understand the details of the study including its aims, methods and use of data.
- 3. I have the right to ask any questions about the study and obtain satisfactory answers from the researchers/doctors.
- 4. I understand that I have the right to withdraw from the study and the healthcare personnel/researchers also have the right to ask my withdrawal due to inappropriate continuation of the study without affecting normal medical care.
- 5. All the information provided by me is correct and will be used for research purposes.
- 6. NTEC-CUHK Cluster REC/IRB will be one of the authorized parties to access the subjects' records related to the study for ethics review purpose.
- 7. I consent to undergo the proposed imaging examinations and further analysis in this study. I understand that magnetic resonance imaging (MRI) are safe imaging modalities, which have been applied in clinical practice for many years. Ultrasound and MRI do not involve ionizing radiation, while only non-ionizing radiation will be produced during scan. The whole process of scanning is

painless. In this study, the standard safety guideline demanded for routine clinical ultrasound and MRI scan will be followed accordingly.

I understand that the subjects undergoing MRI will hear knocking noise resulted from machine running once scan starts, hence ear plugs will be used for hearing protection. Occasionally, the subjects might feel warm because the radiofrequency wave can produce heat.

I understand that, if the subjects feel any uncomfortable or hope to withdraw from ultrasound or MRI examination at any time during scan, they have the right to inform relevant staff to pause scan.

- 8. I consent to use my samples and data for research and/or clinical purposes, which include data acquired from imaging examinations and clinical record.
- 9. To benefit future research, all MRI scans from you will be deposited into the CUHK MRI Data Repository and share with CUHK collaborating partner(s) if necessary. For further analysis of your MRI data, your name will be removed from all scans. Only your gender, age, and disease status (if applied) at the time of scanning will be included.
- 10. I understand and accept that my personal data will be kept for five years after the study.
- 11. I agree that this consent shall remain valid even though the procedures set out in the information sheet may be re-scheduled from time to time.
- 12. I understand that, if I have any further questions, I can contact Dr. H S Leung at (852) 3505-1009 during office hours.
- 13. I understand that, if I have any questions about the ethical issue of this study, I can contact The Joint Chinese University of Hong Kong New Territories East Cluster Clinical Research Ethics Committee at (852) 3505-3935.

| Name | HKID No. |
|-----------|----------|
| Signature | Date |

| I give my informed consent to particip | pate voluntarily in this research | , the above information is true and |
|---|---|---|
| correct to the best of my knowledge. | | |
| Researcher Name: | | |
| Signature: | | |
| Date: | | |